CLINICAL TRIAL: NCT00707655
Title: An Open-label, International, Multi-Center, Phase I/II, Dose-escalation Trial Investigating the Safety of Zalutumumab, a Human Monoclonal Epidermal Growth Factor Receptor Antibody in Combination With Radiotherapy, in Patients With Stage III, IVa or IVb Locally Advanced Squamous Cell Carcinoma of the Head and Neck Ineligible for Platinum Based Chemotherapy
Brief Title: Zalutumumab in Combination With Radiotherapy in Head and Neck Cancer Patients Ineligible for Platinum Based Chemotherapy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The decision is based on company re-evaluation of indications to be pursued within SCCHN
Sponsor: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEN207
Record Dates: First submitted 2008-06-27; First posted 2008-07-01 (Estimated); Results first posted 2011-12-23 (Estimated); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Head and Neck Cancer; Squamous Cell Carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — zalutumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zalutumumab 4 mg/kg (Experimental): Zalutumumab in combination with radiotherapy for 8 weeks. The treatment period of 8 weeks is followed by a 3 week follow-up period where all adverse events are collected and then additionally a 2 year follow-up period where only serious adverse events are collected.
  Interventions: Drug: Zalutumumab
- Zalutumumab 8 mg/kg (Experimental): Zalutumumab in combination with radiotherapy for 8 weeks. The treatment period of 8 weeks is followed by a 3 week follow-up period where all adverse events are collected and then additionally a 2 year follow-up period where only serious adverse events are collected.
  Interventions: Drug: Zalutumumab

INTERVENTIONS:
Drug: Zalutumumab — Eight weekly infusions

SUMMARY:
The purpose of this study is to investigate the safety of zalutumumab in combination with radiotherapy as the treatment of patients with head and neck cancer who are not eligible for platinum based chemotherapy.

DETAILED DESCRIPTION:
This is an open label, multi-center, phase I/II dose-escalation clinical trial investigating the safety of zalutumumab in combination with radiotherapy. The safety of zalutumumab doses in combination with radiotherapy (RT) will be investigated using 3 patient cohorts in a dose-escalation / de-escalation design based on Dose Limiting Toxicity (DLT). The dose-escalation starts at 8 mg/kg zalutumumab in combination with RT. Initially, three patients will be treated at a dose level and observed for DLTs. If none of the three patients experience a DLT, then the next cohort of three patients is treated at the next higher dose of zalutumumab. If one of three patients treated at a dose level experience a DLT, then three more patients are treated at the same dose level. If two or more of the three patients experience DLTs, then the next cohort of three patients should be treated at the next lower dose of zalutumumab, unless at least six patients on that dose have already been dosed. Furthermore, if 1 or fewer DLTs are observed among six patients at a given dose level, then the next cohort of three patients is treated at the next higher dose of zalutumumab. The maximum tolerated dose will be decided by Genmab based on the recommendations made by the IDMC on the basis of their review of the aggregated safety data.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically confirmed diagnosis of locally advanced squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, or larynx stage III, IVa or IVb
2. Measurable disease defined as one or more target lesions according to RECIST based onCT scan or MRI and clinical evaluation
3. Eligible for intended curative radiotherapy
4. Patients considered ineligible for platinum based chemotherapy based on investigator's judgment
5. Age > 18 years
6. Following receipt of verbal and written information about the study, the patient must provide signed informed consent before any study related activity is carried out

Exclusion Criteria:

1. Prior radiotherapy to the head and neck area
2. Prior chemotherapy administered for cancer in the head and neck area
3. Prior targeted therapy (e.g. EGFR antibodies or EGFR inhibitors)
4. Received the following treatments within 4 weeks prior to Visit 2:

   1. Retinoic acid
   2. Other immunosuppressive drugs (e.g. drugs interfering with the functions of T cells, IL-2 or equivalent)
   3. Any non-marketed drug substance
5. Past or current malignancy other than SCCHN, except for:

   * Cervical carcinoma Stage 1B or less
   * Non-invasive basal cell skin carcinoma
   * Squamous cell skin carcinoma
   * Stage 1 or 2 treated prostate cancer with PSA in the normal range for >2 years post treatment
   * Malignant melanoma with a complete response duration of > 10 years
   * Other cancer diagnoses with a complete response duration of > 5 years
6. Metastatic SCCHN disease
7. Chronic or current infectious disease such as, but not limited to, chronic renal infection and tuberculosis
8. Clinically significant cardiac disease including unstable angina, acute myocardial infarction within six months before Visit 1, congestive heart failure, and arrhythmia requiring anti-arrhythmic therapy, with the exception of extra systoles or minor conduction abnormalities
9. Significant concurrent, uncontrolled medical condition including, but not limited to,hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease considered to preclude trial treatment and/or compliance according to the Investigator's opinion, or any other condition preventing therapy according to the Investigator's opinion
10. Known HIV positive
11. Known active hepatitis B and/or hepatitis C
12. Screening laboratory values:

    * Neutrophils < 1.5 x 109/L
    * Platelets < 100 x109/L
    * Hemoglobin < 6 mmol/L
13. Current participation in any other interventional clinical study
14. Patients known or suspected of not being able to comply with a study protocol (e.g. due to alcoholism, drug dependency, or psychological disorder)
15. Known or suspected hypersensitivity to components of the investigational medicinal Product
16. Breast feeding women or women with a positive pregnancy test at screening blood Sample
17. Males not willing to use adequate contraception during study and for 12 months after last dose of zalutumumab or women of childbearing potential not willing to use adequate contraception as hormonal birth control or intrauterine device during study and for 12 months after last dose of zalutumumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-09; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe MAIGON, Principal Investigator — Centre Georges François Leclerc
Locations (8):
- St-Luc University Hospital, Brussels, Belgium
- France (3):
  - Centre Georges-Francois Leclerc Hospital, Dijon
  - Medical Oncology, Outpatient Clinic, Nantes
  - Institut Claudius Regaud Toulouse, Toulouse
- United Kingdom (4):
  - St James's Institute of Oncology, Leeds
  - The Royal Marsden NHS Foundation Trust, London
  - Christie Hospital NHS Foundation Trust, Manchester
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield

RESULTS

PARTICIPANT FLOW:
Groups:
- Zalutumumab 4 mg/kg; Zalutumumab 8 mg/kg: 8 weekly infusions
Period: Overall Study
Arm/Group | Zalutumumab 4 mg/kg | Zalutumumab 8 mg/kg
Started | 3 | 5
Completed | 3 | 3
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zalutumumab 4 mg/kg | Zalutumumab 8 mg/kg | Total
Number analyzed (Participants) | 3 | 5 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 2 | 2
  >=65 years | 3 | 3 | 6
Age, Continuous [Median (Full Range); unit: years] | 73 [72 to 77] | 70 [43 to 81] | 72 [43 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  France | 0 | 4 | 4
  United Kingdom | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: Number of participants with at least one adverse event. All adverse events are collected during 12 weeks and all serious adverse events are collected during 2 years.
Time Frame: From first dose date up to end of the safety follow up period (Up to 2 years)
Population: Analysis set included all 8 participants who were enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Zalutumumab 4 mg/kg | Zalutumumab 8 mg/kg
Number analyzed (Participants) | 3 | 5
Participants | 3 | 5

2. Secondary Outcome: Number of Participants With Best Overall Tumour Response
Description: The Best Overall Tumour Response defined as the best response recorded from the start of treatment until disease progression or recurrence per RECIST criteria. Complete response (CR) defined as the disappearance of all target lesions. Partial response (PR) defined as at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter. Progressive disease (PD) defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started, or the appearance of one or more new lesions since the prior scan. Stable disease (SD) defined as responses not fulfilling CR, PR or PD.
Time Frame: Up to 2 years
Population: Analysis set included all 8 participants who were enrolled in the study. Overall number of participants analyzed are the participants who are available for the assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Zalutumumab 4 mg/kg | Zalutumumab 8 mg/kg
Number analyzed (Participants) | 3 | 4
Participants
  Complete response | 3 | 1
  Partial response | 0 | 3
  Stable disease | 0 | 0
  Progressive disease | 0 | 0

3. Secondary Outcome: Number of Participants With Objective Response
Description: Objective response is defined as CR or PR according to RECIST criteria. CR is defined as the disappearance of all target lesions. PR is defined as at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter.
Time Frame: Up to 2 years
Population: Analysis set included all 8 participants who were enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Zalutumumab 4 mg/kg | Zalutumumab 8 mg/kg
Number analyzed (Participants) | 3 | 5
Participants | 3 | 4

ADVERSE EVENTS:
Time Frame: From first dose date up to end of the safety follow up period (Up to 2 years)
Arm/Group | Zalutumumab 4 mg/kg | Zalutumumab 8 mg/kg
Serious Adverse Events (participants affected / at risk) | 2/3 | 3/5
Other Adverse Events (participants affected / at risk) | 3/3 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zalutumumab 4 mg/kg (N=3) | Zalutumumab 8 mg/kg (N=5)
Oral mucositis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 1 (1)
Loss of weight (Investigations) | 0 (0) | 1 (1)
Mucositis (General disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Disease progression (General disorders) | 0 (0) | 1 (1)
Febrile multifactorial confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zalutumumab 4 mg/kg (N=3) | Zalutumumab 8 mg/kg (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 2 (3)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Disease progression (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 1 (1)
Infusion related reaction (General disorders) | 0 (0) | 1 (1)
Mucosal hemorrhage (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 1 (1) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 2 (2) | 0 (0)
Radiation skin injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Blood magnesium (Investigations) | 0 (0) | 1 (1)
Blood magnesium decreased (Investigations) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1)
Cardiac murmur (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Confusional state (Psychiatric disorders) | 0 (0) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (7)
Skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Mucosal Inflammation (General disorders) | 1 (1) | 5 (7)

LIMITATIONS AND CAVEATS:
All adverse events were collected during the 8 week treatment period and for 4 additional weeks. Serious adverse events were collected for the extended follow-up period of 2 years.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The site and the PI may be required to withhold the publication for up to 90 days. Subject to a reasoned request from the sponsor, the publication may be further delayed for a period up to 6 months from the date of first submission to the sponsor.

The sponsor has the right to require deletion of any trade secret, proprietary, or confidential information supplied by the sponsor to the site or the PI. The sponsor shall not otherwise have the right to censor publications.